CLINICAL TRIAL: NCT02732522
Title: Comparison Between Vaginal and Sublingual Misoprostol 50 µg for Cervical Ripening Prior to Induction of Labor: Randomized Clinical Trial
Brief Title: Comparison Between Vaginal and Sublingual Misoprostol 50 µg for Cervical Ripening Prior to Induction of Labor
Acronym: CMVS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de la Republica (Other)
Responsible Party: Principal Investigator, Andrés Conde, M.D., Universidad de la Republica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMVS-01
Record Dates: First submitted 2016-03-28; First posted 2016-04-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Cervical Ripening
Keywords: misoprostol; induction of labor; sublingual

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol sublingual (Experimental)
  Interventions: Drug: Sublingual misoprostol
- Misoprostol vaginal (Active Comparator)
  Interventions: Drug: Vaginal misoprostol

INTERVENTIONS:
Drug: Sublingual misoprostol
  Arms: Misoprostol sublingual
Drug: Vaginal misoprostol
  Arms: Misoprostol vaginal

SUMMARY:
To analyze whether there is a statistically significant difference in the modifications present in the uterine cervix 6 hours after administration of misoprostol 50 µg through vaginal versus sublingual routes.

DETAILED DESCRIPTION:
A randomized, single blind clinical trial, was performed. Inclusion criteria were all pregnant women admitted at Pereira Rossell Hospital Center with gestational ages between 32/0 and 41/6 according to first trimester sonogram, with a viable fetus in cephalic presentation, with estimated fetal weight lower than 4000 gr, without contraindications for vaginal birth, to whom induction of labor with misoprostol had been previously indicated, from 8 to 20 hours 7 days a week. Protocol counted with approval of the Ethics Commission of the Pereira Rossell Hospital. All participants gave written informed consent before the study began. Once there was confirmation that the patient met the inclusion criteria, information was given and consent form was signed, the patient entered the study and the intervention was randomized. Randomization was computer generated in permuted blocks of 2 by an epidemiologist from our Service, and the result was in a sealed and opaque envelope which was opened at the time of administering the medication. Prior to administration of the medication, an Obstetrician or Obstetrics resident who was not familiar with the administration route assigned to the patient assessed through vaginal examination the characteristics of the cervix in terms of Bishop score. Afterwards, a technician from the investigation team administered the misoprostol according to the assigned route (50 µg misoprostol vaginal or sublingual).

Tachysystole was defined as the presence of at least 6 uterine contractions in 10 minutes.

Primary result was defined as the clinically significant variation (of at least 2 points) of the Bishop score at 6 hours after administration of 50 µg misoprostol. Secondary results were defined as the presence of tachysystole, frequency of vaginal birth and cesarean section, frequency in which new doses were needed to continue with induction of labor and frequency with which labor was diagnosed at 6 hours of administration of misoprostol. Neonatal results included Apgar score at 1 and 5 minutes and pH value in umbilical cord gasometry. Final analysis was made according to intention to treat.

In order to detect a difference in the mean of Bishop score of 2 points, using a standard deviation of 2, with a 90% power, reaching a confidence interval of 95%, a population of 49 patients was required for each group.

Randomization was done in permuted blocks of 2, using a table of randomized numbers. Group 1 included those patients who received sublingual misoprostol and group 2 those patients who received vaginal misoprostol. Analysis was done in statistical package SPSS (reg) V16. For continuous variables a mean and standard deviation were described; for categorical variables absolute frequency and percentage were described. For statistical analysis a 2-tiled independent t-test was used, in order to compare the mean of the two groups. Also, chi-squared test and Fisher´s exact test were used to compare proportions among the two groups where it corresponds.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women admitted at Pereira Rossell Hospital Center
* Gestational ages between 32/0 and 41/6 according to first trimester sonogram
* A viable fetus in cephalic presentation
* Estimated fetal weight lower than 4000 gr
* Without contraindications for vaginal birth
* Whom induction of labor with misoprostol had been previously indicated, from 8 to 20 hours 7 days a week.

Exclusion Criteria:

* Does not meet inclusion criteria.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Bishop score at 6 hours after administration of misoprostol | 6 hours

SECONDARY OUTCOMES:
Number of participants with Tachysystole | 6 hours
  Tachysystole was defined as the presence of at least 6 uterine contractions in 10 minutes.
Number of patients who ended their pregnancy by caesarean section | From administration of misoprostol to birth, up to 3 days.
Requirement of further doses of misoprostol | From administration of misoprostol to birth, up to 3 days.
Labor within 6 hours | 6 hours
Apgar score at 1 minute | At the first minute after delivery
Apgar score at 5 minutes | At the fifth minute after delivery
pH cord blood gas | At delivery

REFERENCES:
- [Derived] Conde A, Ben S, Tarigo J, Artucio S, Varela V, Grimaldi P, Sosa C, Alonso J. Comparison between vaginal and sublingual misoprostol 50 microg for cervical ripening prior to induction of labor: randomized clinical trial. Arch Gynecol Obstet. 2017 Apr;295(4):839-844. doi: 10.1007/s00404-017-4297-9. Epub 2017 Feb 16. PMID 28204882